CLINICAL TRIAL: NCT00555217
Title: CSP #565 - Combination Angiotensin Receptor Blocker and Angiotensin Converting Enzyme Inhibitor for Treatment of Diabetic Nephropathy (VA NEPHRON-D Study)
Brief Title: VA NEPHRON-D: Diabetes iN Nephropathy Study
Acronym: VA NEPHRON-D
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It was stopped primarily because of safety concerns along with low conditional power to detect a treatment effect on the primary outcome.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 565
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Disease; Nephropathy; Type 2 Diabetes
Keywords: kidney disease; nephropathy; type 2 diabetes; hyperkalemia; acute kidney injury
MeSH Terms: conditions — Kidney Diseases; Diabetes Mellitus, Type 2; Hyperkalemia; Acute Kidney Injury | interventions — Losartan; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination of ARB and ACEI (Experimental): Combination of an angiotensin converting enzyme inhibitor (ACEI) with an angiotensin receptor blocker (ARB)
  Interventions: Drug: losartan; Drug: lisinopril
- Monotherapy ARB (Active Comparator): Mono therapy arm. Standard treatment with angiotensin receptor blocker (ARB)
  Interventions: Drug: losartan

INTERVENTIONS:
Drug: losartan — 50 or 100mg/day
Drug: lisinopril — 10, 20 or 40 mg/day
  Arms: Combination of ARB and ACEI

SUMMARY:
Diabetes is the leading cause of end-stage renal disease (ESRD) in the United States. The overall rate of ESRD secondary to diabetes has risen 68% since 1992. Medications that block the renin angiotensin system have been shown to decrease the progression of diabetic nephropathy. The use of an angiotensin receptor blocker (ARB) has been shown to decrease the risk of progression of kidney disease in two studies of individuals with Type 2 diabetes and proteinuria. Despite the use of an ARB, the incidence of renal failure remained high in the treated group in both studies. The combination of an angiotensin converting enzyme inhibitor (ACEI) and ARB can lead to more complete blockade of the renin angiotensin system. In diabetic kidney disease, combination therapy has been shown to decrease proteinuria in short-term studies. Although there are encouraging results for improvement in proteinuria there are no data on progression of kidney disease for the use of combination of ACEI and ARB therapy in patients with diabetes. In addition, there could be an increased risk of serious hyperkalemia in individuals with diabetes who receive combination ACEI and ARB. The investigators therefore propose a randomized double blind multi-center clinical trial to assess the effect of combination of ACEI and ARB in patients with diabetes and proteinuria on progression of kidney disease.

DETAILED DESCRIPTION:
Primary Hypothesis:

To evaluate the combination of an angiotensin converting enzyme inhibitor (ACEI) with an angiotensin receptor blocker (ARB) vs. standard treatment with angiotensin receptor blocker on the progression of kidney disease in individuals with Type 2 diabetes and overt nephropathy.

The primary outcome is a composite endpoint of reduction in estimated GFR of 30 ml/min/1.73m*m in individuals with an estimated baseline GFR greater than or equal to 60 ml/min/1.73m*m; reduction in estimated GFR of greater than 50% in individuals with an estimated baseline GFR less than 60 mL/min/1.73m*m; progression to end-stage renal disease (defined as need for dialysis, renal transplant or an eGFR less than 15 ml/min/1.73m*m) or death.

Secondary outcome: a renal composite endpoint, defined as; reduction in estimated GFR of more than 50% (for individuals with a baseline estimated GFR less than 60 ml/min/1.73m*m); reduction in estimated GFR of more than 30 ml/min/1.73m*m (for individuals with a baseline estimated GFR greater than or equal to 60 ml/min/1.73m*m) or progression to end-stage renal disease (defined as need for dialysis, renal transplant or an eGFR of less than 15 ml/min/1.73m*m).

Tertiary outcomes are cardiovascular events (cardiovascular mortality, myocardial infarction, cerebrovascular accident, admission for heart failure), change in albuminuria at 12 months and decline in slope of kidney function.

Study Abstract:

The study is a multi-center, prospective, randomized, parallel group trial to test the efficacy of the combination of an angiotensin converting enzyme inhibitor (ACEI) with an angiotension receptor blocker (ARB) vs. standard treatment with angiotension receptor blocker on the combined end-point. The primary outcome is a composite endpoint of reduction in estimated GFR of 30 ml/min/1.73m*m in individuals with an estimated GFR greater than or equal to 60 ml/min/1.73m*m; reduction in estimated GFR of greater than 50% in individuals with an estimated GFR less than 60 ml/min/1.73m*m; progression to end-stage renal disease (defined as need for dialysis, renal transplant or en eGFR less than 15 ml/min/1.73m*m)or death. The study population is individuals with type 2 diabetes and overt nephropathy.

Eligible subjects who consent to participate will be randomized into either the combination therapy arm or the mono therapy arm. The randomization will be stratified by site and within sites by baseline albuminuria (< 1 vs. greater than or equal to 1 gram/gram creatinine) and eGFR (< 60 vs. greater than or equal to 60 ml/min/1.73m*m). All participants will receive open label therapy with losartan, an ARB, as standard of care. Patients not treated with an ACEI or ARB will be initiated on losartan; patients treated with an ACEI or ARB other than losartan (the study ARB) will be converted to losartan (the study ARB) and the dose titrated to 100 mg/day. Individuals who tolerate ARB 100mg/day criteria will be randomized in a 1:1 ratio to the addition of blinded lisinopril (the study ACEI) or placebo. The medication (lisinopril or placebo) will be titrated from an initial dose of 10 mg/day to a target dose of 40 mg/day. After each adjustment in dose, serum chemistries will be evaluated for kidney function and potassium levels. Subjects will be enrolled over a period of 4.25 years and the maximum length of follow-up is 6.25 years. The planned study duration is 6.25 years with 4.25 years of accrual and 6.25 years of follow-up for all enrolled patients. The intervention was stopped on November 7, 2012 for safety concerns after an interim analysis. Patients are still under passively follow-up without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Albuminuria >300mg/gram creatinine
* Stage 2 or 3 CKD (eGFR 30 to <90 mg/min/1.73m*2 )
* Able to give informed consent
* Telephone contact available

Exclusion Criteria:

* History of intolerance to ACEI or ARB
* Serum potassium level >5.5 meq/L
* Receiving sodium polystyrene sulfonate (Kayexalate)
* Pregnancy, breast feeding, planning to become pregnant or sexually active and not using birth control
* Renal transplant recipient
* Suspected non-diabetic kidney disease
* Inability to discontinue current use of ACEI/ARB combination
* Current use of Lithium
* Severe (end-stage) comorbid disease
* Prisoner
* Age <18
* Estimated glomerular filtration rate (GFR) <30 or >=90 ml/min/1.73m*m
* HbA1c >10.5%
* Patient refusal
* Participation in a concurrent interventional study
* Blood pressure >180/95
* Unwilling to stop any proscribed medications after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1448 (Actual)
Dates: Start 2008-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Fried, MD MPH, Study Chair — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (31):
- United States (30):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, Little Rock, Arkansas
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - VA Medical Center, Miami, Miami, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - VA Medical Center, St Louis, St Louis, Missouri
  - VA Medical Center, Omaha, Omaha, Nebraska
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Portland, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - WJB Dorn Veterans Hospital, Columbia, Columbia, South Carolina
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA Medical Center, Nashville, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Background] Fried LF, Duckworth W, Zhang JH, O'Connor T, Brophy M, Emanuele N, Huang GD, McCullough PA, Palevsky PM, Seliger S, Warren SR, Peduzzi P; VA NEPHRON-D Investigators. Design of combination angiotensin receptor blocker and angiotensin-converting enzyme inhibitor for treatment of diabetic nephropathy (VA NEPHRON-D). Clin J Am Soc Nephrol. 2009 Feb;4(2):361-8. doi: 10.2215/CJN.03350708. Epub 2008 Dec 31. PMID 19118120
- [Result] Fried LF, Emanuele N, Zhang JH, Brophy M, Conner TA, Duckworth W, Leehey DJ, McCullough PA, O'Connor T, Palevsky PM, Reilly RF, Seliger SL, Warren SR, Watnick S, Peduzzi P, Guarino P; VA NEPHRON-D Investigators. Combined angiotensin inhibition for the treatment of diabetic nephropathy. N Engl J Med. 2013 Nov 14;369(20):1892-903. doi: 10.1056/NEJMoa1303154. Epub 2013 Nov 9. PMID 24206457
- [Result] Fried LF, Emanuele N, Zhang JH. Combined angiotensin inhibition in diabetic nephropathy. N Engl J Med. 2014 Feb 20;370(8):779. doi: 10.1056/NEJMc1315504. No abstract available. PMID 24552328
- [Result] Chen SS, Seliger SL, Fried LF. Complete inhibition of the renin-angiotensin-aldosterone system; where do we stand? Curr Opin Nephrol Hypertens. 2014 Sep;23(5):449-55. doi: 10.1097/MNH.0000000000000043. PMID 25014549
- [Result] Zimering MB, Zhang JH, Guarino PD, Emanuele N, McCullough PA, Fried LF; Investigators for the VA NEPHRON-D. Endothelial cell autoantibodies in predicting declining renal function, end-stage renal disease, or death in adult type 2 diabetic nephropathy. Front Endocrinol (Lausanne). 2014 Aug 11;5:128. doi: 10.3389/fendo.2014.00128. eCollection 2014. PMID 25157242
- [Derived] Tamargo CL, Coca SG, Thiessen Philbrook H, Hu DG, Ix JH, Shlipak MG, Fried LF, Gutierrez OM, Waikar SS, Schrauben SJ, Schelling JR, Ganz P, Kimmel PL, Greenberg JH, Deo R, Takakura A, Vasan RS, Bonventre JV, Parikh CR. The distal nephron biomarkers associate with diabetic kidney disease progression. JCI Insight. 2025 Jun 23;10(12):e186836. doi: 10.1172/jci.insight.186836. eCollection 2025 Jun 23. PMID 40548378
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Huang Y, Fried LF, Kyriakides TC, Johnson GR, Chiu S, Mcdonald L, Zhang JH. Automated safety event monitoring using electronic medical records in a clinical trial setting: Validation study using the VA NEPHRON-D trial. Clin Trials. 2019 Feb;16(1):81-89. doi: 10.1177/1740774518813121. Epub 2018 Nov 16. PMID 30445841

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination of ARB and ACEI | Monotherapy ARB
Started | 724 | 724
Completed | 649 | 656
Not Completed | 75 | 68
Not completed — Withdrawal by Subject | 35 | 31
Not completed — Lost to Follow-up | 19 | 20
Not completed — close out sites | 21 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination of ARB and ACEI | Monotherapy ARB | Total
Number analyzed (Participants) | 724 | 724 | 1448
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.9) | 64.7 (7.7) | 64.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 715 | 721 | 1436
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 75 | 146
  Not Hispanic or Latino | 653 | 649 | 1302
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 25 | 41
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 8 | 5 | 13
  Black or African American | 172 | 160 | 332
  White | 523 | 514 | 1037
  More than one race | 0 | 14 | 14
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 724 | 724 | 1448
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.9 (6.7) | 34.3 (6.9) | 34.6 (6.8)
Coronary Artery Disease [Number; unit: participants]
  Yes | 159 | 167 | 326
  No | 565 | 557 | 1122
Congestive Heart Failure [Number; unit: participants]
  Yes | 116 | 110 | 226
  No | 608 | 614 | 1222
Retinopathy [Number; unit: participants]
  Yes | 309 | 310 | 619
  No | 415 | 414 | 829
SBP [Mean (Standard Deviation); unit: mmHg] | 136.9 (16.5) | 137.0 (16.0) | 136.9 (16.3)
DBP [Mean (Standard Deviation); unit: mmHg] | 72.5 (10.6) | 72.8 (9.9) | 72.7 (10.2)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 157.9 (43.6) | 159.0 (40.5) | 158.4 (42.1)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dl] | 81.6 (32.4) | 84.3 (35.0) | 82.9 (33.7)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dl] | 37.7 (11.0) | 38.7 (11.3) | 38.2 (11.2)
Triglycerides [Median (Inter-Quartile Range); unit: mg/dl] | 165 [111 to 260] | 162 [111 to 235] | 163 [111 to 249]
HbA1c [Mean (Standard Deviation); unit: %] | 7.8 (1.2) | 7.8 (1.3) | 7.8 (1.3)
serum Creatinine at enrollment [Mean (Standard Deviation); unit: mg/dl] | 1.5 (0.4) | 1.5 (0.4) | 1.5 (0.4)
Potassium [Mean (Standard Deviation); unit: meq/L] | 4.3 (0.5) | 4.3 (0.5) | 4.3 (0.5)
eGFR at enrollment [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 53.6 (15.5) | 53.7 (16.2) | 53.7 (15.9)
urine albumin/creatinine at enrollment [Median (Inter-Quartile Range); unit: mg/g] | 841.5 [495 to 1698] | 861.5 [487.5 to 1789] | 851.0 [490 to 1752]

OUTCOME MEASURES:

1. Primary Outcome: A Composite Endpoint of Reduction in Estimated GFR of 30ml/Min/1.73m*m in Individuals w/a Baseline Estimated GFR >= 60 ml/Min/1.73m*m, Reduction in Estimated GFR >50% in Individuals w/ Baseline Estimated GFR <60ml/Min/1.73m*m; ESRD or Death
Description: Time to the first event of reduction in estimated GFR of 30ml/min/1.73m*m in individuals w/a baseline estimated GFR >= 60 ml/min/1.73m*m, reduction in estimated GFR >50% in individuals w/ baseline estimated GFR <60ml/min/1.73m*m; ESRD or death.
Time Frame: From enrollemnt to time of first primary event, up to 4.5 years
Measure: Number; unit: participants
Arm/Group | Combination of ARB and ACEI | Monotherapy ARB
Number analyzed (Participants) | 724 | 724
participants | 132 | 152
Statistical Analysis 1: Comparison: Combination of ARB and ACEI vs Monotherapy ARB; Test type: Superiority or Other; p = 0.30, Log Rank; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.70 to 1.12] — Combination ARB and ACEI vs. mono therapy ARB

2. Secondary Outcome: A Renal Composite Endpoint, Defined as; Reduction in Estimated GFR of >50% (for Individuals With Baseline GFR <60) or Reduction in GFR of >30 (for Individuals With Baseline GFR >= GFR 60) or ESRD.
Description: Time to the first event of reduction in estimated GFR of >50% (for individuals with baseline GFR <60) or reduction in GFR of >30 (for individuals with baseline GFR >= GFR 60) or ESRD.
Time Frame: From enrollment to time of first event, up to 4.5 years
Measure: Number; unit: participants
Arm/Group | Combination of ARB and ACEI | Monotherapy ARB
Number analyzed (Participants) | 724 | 724
participants | 77 | 101
Statistical Analysis 1: Comparison: Combination of ARB and ACEI vs Monotherapy ARB; Test type: Superiority or Other; p = 0.10, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.58 to 1.05] — Combination ARB and ACEI vs. mono therapy ARB

ADVERSE EVENTS:
Time Frame: July 2008 - January 2013
Arm/Group | Combination of ARB and ACEI | Monotherapy ARB
Serious Adverse Events (participants affected / at risk) | 416/724 | 380/724
Other Adverse Events (participants affected / at risk) | 0/724 | 0/724
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of ARB and ACEI (N=724) | Monotherapy ARB (N=724)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 15 (23) | 12 (13)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic pu (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (3) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Normochromic normocytic anaemi (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 7 (8)
Acute myocardial infarction (Cardiac disorders) | 27 (31) | 24 (25)
Angina pectoris (Cardiac disorders) | 7 (8) | 9 (11)
Angina unstable (Cardiac disorders) | 4 (4) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 13 (18) | 14 (19)
Atrial flutter (Cardiac disorders) | 5 (5) | 3 (3)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complet (Cardiac disorders) | 3 (3) | 4 (4)
Atrioventricular block first d (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 8 (8) | 6 (6)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 7 (8) | 6 (6)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 3 (4)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 80 (143) | 95 (155)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (3) | 2 (2)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 32 (35) | 23 (26)
Coronary artery occlusion (Cardiac disorders) | 6 (7) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 7 (7) | 7 (7)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 18 (18) | 15 (17)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Nodal rhythm (Cardiac disorders) | 2 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (3)
Rhythm idioventricular (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 2 (2) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Trifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Haemorrhagic arteriovenous mal (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemor (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 14 (17) | 5 (5)
Gastrointestinal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorr (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (5) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Lower gastrointestinal haemorr (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 2 (4)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 2 (2)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (7) | 2 (4)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorr (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Adverse drug reaction (General disorders) | 4 (5) | 2 (2)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 3 (3)
Chest pain (General disorders) | 24 (27) | 21 (26)
Death (General disorders) | 25 (25) | 13 (13)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Hernia obstructive (General disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (2)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Medical device complication (General disorders) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 7 (7) | 6 (6)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 4 (4)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 4 (4) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 33 (46) | 31 (39)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 6 (6) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 2 (2) | 0 (0)
External ear cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 6 (7) | 4 (5)
Gastroenteritis (Infections and infestations) | 9 (10) | 4 (4)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 3 (3)
Graft infection (Infections and infestations) | 1 (1) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 3 (4) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 6 (6) | 5 (5)
Localised infection (Infections and infestations) | 2 (3) | 1 (1)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 13 (17) | 13 (15)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Peptostreptococcus infection (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 43 (50) | 41 (43)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 3 (3) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 3 (3)
Sepsis syndrome (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (2) | 2 (2)
Staphylococcal infection (Infections and infestations) | 6 (6) | 4 (4)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Subdural empyema (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infect (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 14 (16) | 9 (10)
Urosepsis (Infections and infestations) | 3 (3) | 2 (2)
Viral cardiomyopathy (Infections and infestations) | 0 (0) | 1 (1)
West Nile viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 4 (5) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site com (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Arteriovenous fistula thrombos (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 17 (18) | 20 (22)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
In-stent coronary artery reste (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complicati (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation dysphagia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 9 (11)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Antibiotic resistant Staphyloc (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level abo (Investigations) | 1 (1) | 1 (1)
Anticoagulation drug level bel (Investigations) | 1 (1) | 0 (0)
Biopsy kidney (Investigations) | 0 (0) | 2 (2)
Biopsy lung (Investigations) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase i (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 3 (3)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram change (Investigations) | 1 (1) | 0 (0)
Fistulogram (Investigations) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
International normalised ratio (Investigations) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Diabetes mellitus inadequate c (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (3)
Fluid overload (Metabolism and nutrition disorders) | 7 (12) | 6 (6)
Gout (Metabolism and nutrition disorders) | 5 (6) | 6 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (10) | 16 (16)
Hyperglycaemic hyperosmolar no (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 39 (45) | 16 (16)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 19 (21) | 20 (27)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degenerati (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (8)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (6)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (8) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung squamous cell carcinoma s (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nasopharyngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma of th (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma metastati (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer stage u (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic nervous system imbal (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 2 (2) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (3) | 4 (4)
Central nervous system mass (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 3 (3) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 12 (12) | 10 (12)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (3) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 10 (10) | 9 (10)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 5 (5) | 10 (12)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Drug abuse (Psychiatric disorders) | 4 (4) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 5 (5) | 6 (6)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 9 (10) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (3)
Azotaemia (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic end stage renal disea (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (3) | 2 (4)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 3 (3)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 5 (6)
Renal failure acute (Renal and urinary disorders) | 130 (190) | 80 (105)
Renal failure chronic (Renal and urinary disorders) | 4 (5) | 7 (7)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 3 (3)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 3 (3)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 14 (20) | 22 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 4 (5)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (7)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 7 (8) | 10 (12)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (5)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Treatment noncompliance (Social circumstances) | 5 (5) | 4 (4)
Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous fistula operatio (Surgical and medical procedures) | 2 (2) | 1 (3)
Arthrotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Brachytherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary arterial stent insert (Surgical and medical procedures) | 1 (1) | 4 (4)
Coronary artery bypass (Surgical and medical procedures) | 2 (2) | 0 (0)
Drug rehabilitation (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Ethmoid sinus surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Extubation (Surgical and medical procedures) | 0 (0) | 1 (1)
Foot amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric banding (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrointestinal tube insertio (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemodialysis (Surgical and medical procedures) | 2 (2) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Leg amputation (Surgical and medical procedures) | 2 (2) | 0 (0)
Penile prosthesis insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Therapy regimen changed (Surgical and medical procedures) | 1 (1) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 2 (2) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 2 (3) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 6 (6)
Hypertensive crisis (Vascular disorders) | 4 (4) | 4 (4)
Hypertensive emergency (Vascular disorders) | 3 (3) | 3 (4)
Hypotension (Vascular disorders) | 11 (13) | 8 (8)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (3) | 6 (6)
Peripheral arterial occlusive (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 3 (3) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 4 (6) | 3 (3)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Thrombosed varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
In October, 2012 the DMC recommended that study treatment be stopped primarily because of safety concerns along with low conditional power to detect a treatment effect on the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No